CLINICAL TRIAL: NCT03552900
Title: Evaluating the Use of a Mobile App to Reduce Symptoms of Depression and Anxiety for Students Seeking Care at Harvard University Health Services
Brief Title: Evaluating a Mobile App for Students Seeking Care for Depression and Anxiety at Harvard University Health Services
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harvard University (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Leslie Tarver, Physician Researcher, Harvard University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB17-1876
Record Dates: First submitted 2018-03-27; First posted 2018-06-12 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Depression, Anxiety
MeSH Terms: conditions — Depression; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two study groups and assigned to one of two different mobile apps
Who Masked: Investigator
Masking Description: Participants will not be masked to their mobile app however investigators conducting data analysis will be blinded to which participants were assigned to which app
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- App 1 Study group (7cups) (Active Comparator): Participants assigned to this group will be assigned a behavioral intervention, the mobile app ("7cups") which allows participants access to direct online social support via the app.
  Interventions: Behavioral: 7cups Mobile App
- App 2 Study Group (Bliss (Active Comparator): Participants assigned to this group will be assigned to a behavioral intervention, the mobile app (" Bliss ") which provides participants an informational app about mental health resources at Harvard.
  Interventions: Behavioral: Bliss

INTERVENTIONS:
Behavioral: 7cups Mobile App — Participants who receive the 7 Cups mobile app will get access to direct online social support by messaging with a listener, participating in group chats as well as evidence-based information and exercises to promote their mental health.
  Arms: App 1 Study group (7cups)
Behavioral: Bliss — Participants who receive the Bliss app will get access to an app that that provides access to important community, health, wellness, academic, and support resources.
  Arms: App 2 Study Group (Bliss

SUMMARY:
Brief Summary:

Background:

There is a growing demand for mental health services on college campuses. At the same time there has been a dramatic surge in development of mobile mental health apps. Given the widespread popularity and utilization of mobile apps in the college-age population, there is an opportunity to leverage these tools to improve services. The study aims to evaluate the effects of a mobile app on reducing symptoms of depression and anxiety for students awaiting their first visit at Harvard Counseling and Mental Health Services (CAMHS), and on enhancing recovery after beginning treatment.

Methods:

Students seeking an appointment at Harvard CAMHS who meet eligibility criteria will be randomized to receive one of two apps: a direct online social support (7cups) or an app that provides information about community, health, wellness, academic, and support resources on campus (Bliss). Participants will complete a baseline assessment using the PHQ-9 and GAD-7 and a measure of perceived social support. They will be asked to use their assigned app while awaiting their intake appointment and during treatment. The primary endpoint will be at 2 weeks after enrollment and the secondary endpoints at 4, 8- and 12 weeks after enrollment. At all endpoints participants will complete a PHQ-9, GAD-7 and a survey assessing their experience with the app. At the 8-week endpoint they will also be asked about their overall satisfaction with their care and their perceived social support.

Results:

Feasibility and acceptability of the app will be evaluated by analyzing usage metrics of the 7cups app, self-report satisfaction questionnaire as well as trial adherence. Changes in PHQ-9 and GAD-7 scores between the two groups at baseline, primary and secondary endpoints will be analyzed as well as associations between PHQ-9, GAD-7 scores and patient socio-demographic and social support variables. Mediators of change in symptoms including frequency of use, activities used on app and perceived social support will also be analyzed.

DETAILED DESCRIPTION:
Abstract:

There is a growing demand for mental health services on college campuses. At the same time there has been a dramatic surge in development of mobile apps for mental health. Given the widespread popularity and utilization of mobile apps in the college-age population, there is an opportunity to leverage these tools to improve services. The study aims to evaluate the effects of a mobile mental health app on reducing symptoms of depression and anxiety for students awaiting their first visit at Harvard Counseling and Mental Health Services (CAMHS), and Harvard graduate students who have been recommended to seek treatment at CAMHS. The feasibility and acceptability of a mobile app intervention with this population will also be assessed, as well as the ways through which the mobile app may contribute to improvement in depression and anxiety among students such as change in perceived social support for students using a mobile social support app.

Specific Aims:

Untreated or under-treated depression and anxiety in college-age students has tremendous costs for the individual, the larger community and society at large, with the worst, fatal outcome of suicide leading to devastating consequences for college communities. 64% of young adults who are no longer in college are not attending college because of a mental health related condition and the frequency that students in treatment report having "seriously considered suicide" has increased by almost 40% in the last five years. Despite these facts, still only 25% of students with a mental health concern seek treatment. Technological innovations such as mobile apps hold promise to improve access to care, de-stigmatize treatment and potentially alleviate demand on over-burdened service centers. However, there is limited evidence on the effectiveness and feasibility of use of these mobile platforms. Consequently, there is a pressing need to develop better research modalities for evaluating mobile apps and to elucidate the specific features that are effective at reducing symptoms and are acceptable in this population in order to improve care and inform novel treatment approaches.

In this study, participants seeking mental health services at a university health center will receive a mobile social support app. The investigators hypothesize that receiving immediate access to a mobile, anonymous social support app while waiting for an appointment and during treatment will be feasible and acceptable to young adults seeking mental health services, and will yield promising results for improving outcomes of depression and anxiety in comparison to those in the control group. The pilot deign will address the following aims:

Aim1: Evaluate the potential effectiveness of a mobile social support app at reducing symptoms of depression and anxiety for students seeking mental health services.

Aim 2: Assess the feasibility and acceptability of providing students access to a mobile social support app to augment available mental health services within a university health center.

Aim 3: Test the feasibility of conducting a fully remote, digital trial with college students seeking mental health services with randomization to a mobile social support app.

Background and Significance:

There is a mental health crisis on college campuses across the country. 64% of young adults who are no longer in college are not attending college because of a mental health related condition and the frequency that students in treatment report having "seriously considered suicide" has increased by almost 40% in the last five years. The demand for counseling services has also grown at least five times faster than average student enrollment. This has led to a significant shortage of mental health services for students.

Considering the ubiquity of mobile phone usage, particularly in this population -over 86% of young adults aged 18-29 owns a smart phone-there is significant interest in the use of mobile phone apps as a powerful alternate care delivery platform. Additionally, the number of mobile mental health apps is exponentially growing with currently thousands of mental health apps available for download on the Apple or Google Marketplaces. Given their widespread use, mobile apps have the potential to reach people outside of the traditional care model and allow people to use these tools when they need them, and as often as they like without having to wait for a mental health professional.

There are numerous potential advantages of mobile health applications, such as continuous availability and immediate support, anonymity, customizable content and self-guided treatment approaches. Additionally, these approaches hold promise for increasing access to care particularly for those in remote areas and traditionally hard-to-reach groups. These tools have also been seen as ways to increase service capacity and efficiency, reduce other barriers to face-to-face help seeking such as stigma and shame, and may be particularly well suited to young people who may be more accepting of technological approaches.

However, despite the growing number of apps available and the consensus that these innovations hold promise for expanding mental health care delivery, the evidence base for their efficacy remains unclear and research is significantly lagging behind app development. A review of mHealth apps for the most prevalent conditions identified by the WHO identified more than 1536 apps for depression, but only 32 associated published articles. Many mobile platforms developed by commercial companies are widely utilized but have not been adequately evaluated to determine their effectiveness. In a scoping review of the literature on mobile apps for mental health in adolescents, only two RCTs were identified and both failed to demonstrate a significant effect on intended outcomes. A large meta-analysis conducted recently on smartphone interventions for depressive symptoms in adults found a moderate positive effect on depressive symptoms, however, the subgroup analyses found that the effects of smart- phone interventions were substantially larger when compared to inactive (g= 0.56) than active (g=0.22) control conditions.

Further, there is a broad spectrum of features ranging from entirely self-guided tools, mixed approaches that combine self-guided tools with interactions with coaches or fully structured programs with an therapist or coach guiding treatment. There is a lack of evidence, however, about which features are most helpful and which approach is best suited for an individual or given population. The evidence on self-guided alone versus provider-supported internet based treatments does indicate that human support significant improves engagement. Initial study findings and high drop out rates also suggests that a major challenge with mobile apps is user attrition and decreased engagement over time. This is where human connection and social support features may play a critical role in maintaining interest and engagement. This pilot study aims to contribute to the understanding of the use of mobile mental health apps targeting a college-age population. By selecting a mainly social support app, it also aims to explore to what degree enhanced social support plays a role in improved outcomes.

Research Design:

This is a pilot study evaluating the acceptability and outcomes of a mobile social support app, 7 cups which is commercially available and widely utilized by the target population, to reduce symptoms of depression and anxiety for college students seeking mental health services and selected graduate students who have completed a mental health screening and are recommended to seek treatment at CAMHS..

Methods

Recruitment and Screening:

When students make an initial consultation appointment online for counseling and mental health services (CAMHS), they will be able to click a link about the study which directs them to the study enrollment website. Interested participants will complete a survey to determine eligibility including information about basic demographics and mobile device ownership. Those meeting basic eligibility requirements will also complete screening using the Patient Health Questionnaire - 9 and the Generalized Anxiety Disorder 7-item scale to determine final eligibility. If deemed to be eligible, participants will sign an electronic consent form.

Harvard graduate students who have completed a mental wellness survey as part of another research study led by Dr. Barreira, would be invited to participate in this study after completing the survey. For these graduate students, after they complete the survey, if their score indicates mild symptoms of depression or anxiety or greater they would be offered to participate in the mobile app study. It is currently standard practice for graduate students completing the mental wellness surveys that recommendations to seek care at HUHS CAMHS are given If they score with symptoms of depression or anxiety. With the addition of this study, students would now also be invited to participate in the mobile app study as an additional tool to manage their mental and emotional health.

Approximately 500 students present to CAMHS seeking services each month depending on the time of year. We have learned from the pilot study that we are likely to enroll approximately 30% of these students with approximately 30% drop out rate. Additionally, there are approximately 300 Harvard graduate students who have completed a mental health screening and would be invited to participate in the study. Again assuming approximately 30-40% of those students enroll in the study and a 30% drop out rate. Thus we anticipate obtaining usable data from approximately 150 participants. This sample size would allow us to obtain 0.80 power to detect significant improvement (Cohen d = 0.4) assuming significance 0.05.

Baseline Assessment and Group Assignment:

Once enrolled, participants will be asked additional questions to provide baseline assessment such as brief additional demographic information which will include participants' class year, race/ethnicity, use of other mental health apps, and current engagement in mental health treatment. We will ask participants for an email address and phone number for study staff to be able to contact them during the study. In addition, participants will be asked about current use of substances or alcohol as this is known to affect treatment outcomes. This will be collected using the AUDIT-C, a 3-item alcohol screen, which is a modified version of the 10-question AUDIT instrument. Participants will also be asked to complete a brief set of questions about perceived social support to obtain a baseline assessment using the Multidimensional Scale of Perceived Social Support. Participants will then be randomly assigned to one of two apps: an app offering direct online social support (7cups) or an app that provides information about mental health resources on campus (Bliss). Following this, participants are guided through the process of downloading their assigned app on their smartphone, given instructions on how to reach HUHS urgent care if their symptoms worsen and how to contact the study staff with questions.

ELIGIBILITY:
Inclusion Criteria:

Participants will be required to be Harvard students, 18 years old or older, own a smartphone with Wi-Fi or 3G/4G capabilities and have a triage appointment scheduled with Harvard Counseling and Mental Health. Those meeting basic eligibility requirements will also complete screening using the Patient Health Questionnaire - 9 and the Generalized Anxiety Disorder 7-item scale to determine final eligibility and obtain baseline assessment. A PHQ-9 score of 5 or greater, or a score of 2 or greater on PHQ item 10 (indicating that they felt disabled in their life because of their mood) or a GAD-7 score of 8 or greater will be required for enrollment.

Exclusion Criteria: Those who score less than 5 on PHQ-9 or less than 8 on the GAD-7 during study screening will be excluded from the study and sent an automated message with information to contact HUHS CAMHS if their symptoms worsen and they need to be seen urgently.

*Participants with a PHQ-9 suicide item score of 1 or more will not be excluded from the study but will receive an automated message with information to call HUHS urgent care if they are feeling at risk of harm to themselves or others. Study staff will also notify CAMHS staff within one business day so that a member of staff can reach out to the participant and check in about scheduling an urgent care appointment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-04-16 (Actual); Primary Completion 2018-07-16 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
Patient Health Questionnaire - 9 (PHQ-9) | At two weeks after enrollment, participants will receive an email to complete the PHQ-9 and GAD-7, which will serve as the primary outcome measure of the study.
  The PHQ-9 is a 9-question multipurpose instrument for screening, diagnosing, monitoring and measuring the severity of depression.
  The Patient Health Questionnaire (PHQ-9) Scoring:
  Scoring: 0-3 Scale for each item; 0 Not at all; 3 Nearly every day
  The nine item version of the Patient Health Questionnaire (PHQ-9) was designed to facilitate the recognition and diagnosis of depression in primary care patients. It can be used to monitor change in symptoms over time and provides a depression severity index score as follows:
  0-4 None 5-9 Mild 10 - 14 Moderate 15 - 19 Moderately Severe 20 - 27 Severe
  The recommended cut-off for the PHQ-9 severity index is a score of 9. Anyone who scores 10 or above can be considered to be suffering from clinically signicant symptoms of depression.
Generalized Anxiety Disorder 7-item scale (GAD-7) | At two weeks after enrollment, participants will receive an email to complete the PHQ-9 and GAD-7, which will serve as the primary outcome measure of the study.
  The GAD-7 is a 7 item instrument for screening and severity measuring of generalized anxiety disorder (GAD).
  Scoring: 0-3 Scale for each item; 0 Not at all; 3 Nearly every day
  The index scores are as follows:
  0-4 None 5-10 Mild Anxiety 11 - 15 Moderate Anxiety 15 - 21 Severe Anxiety
  The recommended cut off for the GAD-7 severity index is a score of 7. Anyone who scores 8 or above can be considered to be suffering from clinically significant anxiety symptoms.

SECONDARY OUTCOMES:
Multidimensional Scale of Perceived Social Support | Participants will receive this instrument at baseline, and at the 4 and 8-week endpoint.
  Instrument to assess participant's perceived social support. Includes 12 questions where participants rate their responses on a scale of 1 to 7 ("1" Very Strongly Disagree, "2" Strongly Disagree, "3" Mildly Disagree, "4" Neutral, "5" Mildly Agree, "6" Strongly Agree "7" Very Strongly Agree).
  The items can be divided into subgroups relating to the source of social support, namely family (Fam), friends (Fri) or significant other (SO).
  Scoring Information: To calculate mean scores:
  Significant Other Subscale: Sum across items 1, 2, 5, & 10, then divide by 4. Family Subscale: Sum across items 3, 4, 8, & 11, then divide by 4. Friends Subscale: Sum across items 6, 7, 9, & 12, then divide by 4. Total Scale: Sum across all 12 items, then divide by 12.
  The 12-item MSPSS scale has a mean continuous score ranging from 1-84. Higher scores indicate greater perceived social support.
Client Satisfaction Questionnaire (CSQ-8) | Participants will receive a survey to complete this questionnaire at the 8 week endpoint
  Questionnaire to assess patient satisfaction with care.
  The CSQ-8 is a brief measure to assess patients' satisfaction the service they received from university health services. CSQ-8 is an 8-item scale with scores that range from 8 to 32, with higher values indicating higher satisfaction.
Participant Experience Survey | Participants will receive a survey to complete this questionnaire at the 2, 4, 8 and 12 week endpoint
  12-item questionnaire to measure participant's qualitative experiences with their assigned mobile app including overall utility, what activities were most used, help achieving goals, etc.
Secondary Process Outcome Survey | Participants will receive a survey to complete this questionnaire at the 4 and 8 week endpoint
  4 items to assess participants' use of other forms of care during the study including urgent mental health care, primary care and seeking help from others

CONTACTS AND LOCATIONS:
Overall Officials: Leslie Tarver, MD, Principal Investigator — Harvard University; Paul Barreira, MD, Study Director — Harvard University
Locations (1):
- Harvard University Health Services, Cambridge, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Aboujaoude E, Salame W, Naim L. Telemental health: A status update. World Psychiatry. 2015 Jun;14(2):223-30. doi: 10.1002/wps.20218. PMID 26043340
- [Background] Van Ameringen M, Turna J, Khalesi Z, Pullia K, Patterson B. There is an app for that! The current state of mobile applications (apps) for DSM-5 obsessive-compulsive disorder, posttraumatic stress disorder, anxiety and mood disorders. Depress Anxiety. 2017 Jun;34(6):526-539. doi: 10.1002/da.22657. Epub 2017 Jun 1. PMID 28569409
- [Background] American College Health Assocation. American College Health Association-National College Health Assessment II: Reference Group Executive Summary Spring 2013. Linthicum, MD: American College Health Association; 2013.
- [Background] Anderson M. Technology device ownership. Washington, DC: Pew Research Center; 2015.
- [Background] Arean PA, Hallgren KA, Jordan JT, Gazzaley A, Atkins DC, Heagerty PJ, Anguera JA. The Use and Effectiveness of Mobile Apps for Depression: Results From a Fully Remote Clinical Trial. J Med Internet Res. 2016 Dec 20;18(12):e330. doi: 10.2196/jmir.6482. PMID 27998876
- [Background] Baumel A. Online emotional support delivered by trained volunteers: users' satisfaction and their perception of the service compared to psychotherapy. J Ment Health. 2015;24(5):313-20. doi: 10.3109/09638237.2015.1079308. PMID 26485198
- [Background] Blanco C, Okuda M, Wright C, Hasin DS, Grant BF, Liu SM, Olfson M. Mental health of college students and their non-college-attending peers: results from the National Epidemiologic Study on Alcohol and Related Conditions. Arch Gen Psychiatry. 2008 Dec;65(12):1429-37. doi: 10.1001/archpsyc.65.12.1429. PMID 19047530
- [Background] Broglia E, Millings A, Barkham M. Comparing counselling alone versus counselling supplemented with guided use of a well-being app for university students experiencing anxiety or depression (CASELOAD): protocol for a feasibility trial. Pilot Feasibility Stud. 2017 Jan 23;3:3. doi: 10.1186/s40814-016-0119-2. eCollection 2017. PMID 28127442
- [Background] Center for Collegiate Mental Health (CCMH). 2015 Annual Report. Publication No. STA 15-108. January 2016. https://sites.psu.edu/ccmh/files/2017/10/2015_CCMH_Report_1-18-2015-yq3vik.pdf
- [Background] Center for Collegiate Mental Health (CCMH). 2016 Annual Report. Publication No. STA 17-74. January, 2017. <https://sites.psu.edu/ccmh/files/2017/01/2016-Annual-Report-FINAL_2016_01_09-1gc2hj6.pdf>
- [Background] Fairburn CG, Patel V. The impact of digital technology on psychological treatments and their dissemination. Behav Res Ther. 2017 Jan;88:19-25. doi: 10.1016/j.brat.2016.08.012. PMID 28110672
- [Background] Firth J, Torous J, Nicholas J, Carney R, Pratap A, Rosenbaum S, Sarris J. The efficacy of smartphone-based mental health interventions for depressive symptoms: a meta-analysis of randomized controlled trials. World Psychiatry. 2017 Oct;16(3):287-298. doi: 10.1002/wps.20472. PMID 28941113
- [Background] Grist R, Porter J, Stallard P. Mental Health Mobile Apps for Preadolescents and Adolescents: A Systematic Review. J Med Internet Res. 2017 May 25;19(5):e176. doi: 10.2196/jmir.7332. PMID 28546138
- [Background] Gruttadaro, D and Crudo D., National Alliance on Mental Illness: College Students Speak: A Survey Report on Mental Health. 2012.
- [Background] Kauer SD, Reid SC, Crooke AH, Khor A, Hearps SJ, Jorm AF, Sanci L, Patton G. Self-monitoring using mobile phones in the early stages of adolescent depression: randomized controlled trial. J Med Internet Res. 2012 Jun 25;14(3):e67. doi: 10.2196/jmir.1858. PMID 22732135
- [Background] Kenny R, Dooley B, Fitzgerald A. Developing mental health mobile apps: Exploring adolescents' perspectives. Health Informatics J. 2016 Jun;22(2):265-75. doi: 10.1177/1460458214555041. Epub 2014 Nov 10. PMID 25385165
- [Background] Larsen DL, Attkisson CC, Hargreaves WA, Nguyen TD. Assessment of client/patient satisfaction: development of a general scale. Eval Program Plann. 1979;2(3):197-207. doi: 10.1016/0149-7189(79)90094-6. No abstract available. PMID 10245370
- [Background] Marzano L, Bardill A, Fields B, Herd K, Veale D, Grey N, Moran P. The application of mHealth to mental health: opportunities and challenges. Lancet Psychiatry. 2015 Oct;2(10):942-8. doi: 10.1016/S2215-0366(15)00268-0. Epub 2015 Sep 29. PMID 26462228
- [Background] Mistler, B., et. al. Association for University and College Counseling Center Directors Annual Survey, 2012.
- [Background] Mohr DC, Burns MN, Schueller SM, Clarke G, Klinkman M. Behavioral intervention technologies: evidence review and recommendations for future research in mental health. Gen Hosp Psychiatry. 2013 Jul-Aug;35(4):332-8. doi: 10.1016/j.genhosppsych.2013.03.008. Epub 2013 May 8. PMID 23664503
- [Background] Mohr DC, Tomasino KN, Lattie EG, Palac HL, Kwasny MJ, Weingardt K, Karr CJ, Kaiser SM, Rossom RC, Bardsley LR, Caccamo L, Stiles-Shields C, Schueller SM. IntelliCare: An Eclectic, Skills-Based App Suite for the Treatment of Depression and Anxiety. J Med Internet Res. 2017 Jan 5;19(1):e10. doi: 10.2196/jmir.6645. PMID 28057609
- [Background] Olff M. Mobile mental health: a challenging research agenda. Eur J Psychotraumatol. 2015 May 19;6:27882. doi: 10.3402/ejpt.v6.27882. eCollection 2015. PMID 25994025
- [Background] Schlosser DA, Campellone TR, Truong B, Anguera JA, Vergani S, Vinogradov S, Arean P. The feasibility, acceptability, and outcomes of PRIME-D: A novel mobile intervention treatment for depression. Depress Anxiety. 2017 Jun;34(6):546-554. doi: 10.1002/da.22624. Epub 2017 Apr 18. PMID 28419621
- [Background] Spitzer RL, Kroenke K, Williams JB, Lowe B. A brief measure for assessing generalized anxiety disorder: the GAD-7. Arch Intern Med. 2006 May 22;166(10):1092-7. doi: 10.1001/archinte.166.10.1092. PMID 16717171
- [Background] Sucala M, Cuijpers P, Muench F, Cardos R, Soflau R, Dobrean A, Achimas-Cadariu P, David D. Anxiety: There is an app for that. A systematic review of anxiety apps. Depress Anxiety. 2017 Jun;34(6):518-525. doi: 10.1002/da.22654. Epub 2017 May 15. PMID 28504859
- [Background] Torous J, Roberts LW. The Ethical Use of Mobile Health Technology in Clinical Psychiatry. J Nerv Ment Dis. 2017 Jan;205(1):4-8. doi: 10.1097/NMD.0000000000000596. PMID 28005647